CLINICAL TRIAL: NCT00020722
Title: Treatment of Stage IV Breast Cancer With Activated T Cells After Peripheral Blood Stem Cell Transplant (Pilot Phase II)
Brief Title: Chemotherapy Followed by Peripheral Stem Cell Transplantation Plus Biological Therapy in Treating Women With Stage IV Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding to continue study.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lawrence Lum, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068707; P30CA022453 (NIH); WSU-2007-033 (Other: MI172); RWMC-0634246 (Other: MI172)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ifosfamide; Carboplatin; Etoposide; Ice; Clinical Protocols; etoposide phosphate; Cyclophosphamide; Thiotepa; Leukapheresis; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- therapeutic autologous lymphocytes (Experimental)
  Interventions: Biological: therapeutic autologous lymphocytes; Drug: Ifosfamide, carboplatin, and etoposide (ICE) regimen; Drug: Cyclophosphamide, Thiotepa, Carboplatin (CTC) or STAMP V (CTC); Procedure: Leukapheresis; Procedure: peripheral blood stem cell transplantation (PBSCT)

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes — Immediately after pheresis, the lymphocytes will be activated with soluble monoclonal anti-CD3 antibody (OKT3) which cross-links the CD3 receptors on T cells and activates T cells.
  The time for ATC infusions will vary from patient to patient, but the infusion rate will be based on the rate calculated from the endotoxin level in the cell product. All patients will be observed for at least 1 hr after an infusion.
Drug: Ifosfamide, carboplatin, and etoposide (ICE) regimen — Ifosfamide 2,500 mg/m2 given IV daily on day -8, -7, -6, -5, -4, and -3 prior to PBSCT. Ifosfamide 2,500 mg/m2 infused IV over 1 hour (hour 0-1) on days -8 to -3 for a total dose of 15,000 mg/m2.
  Mesna will be administered per BMT Standard of Care Guideline at a dose of 25% of the total Ifosfamide dose 30 minutes prior to and then 3, 6, and 9 hours after ifosfamide daily on days -8, -7, -6, -5, -4, and -3 prior to PBSCT for a total dose of 2500 mg/m2.
  Carboplatin at a dose of 250 mg/m2 will be given daily on days -8, -7, -6, -5, -4, and -3 prior to PBSCT for a total dose of 1500 mg/m2.
  VP-16 (etoposide) at a dose of 200 mg/m2 will be given IV on days -8, -7, -6, -5, -4 and -3. The total dose of VP-16 given prior to PBSCT will be 2,400 mg/m2. VP-16 will be given 200 mg/m2
  Other Names: Ifex®; Paraplatin ®; Toposar®; VePesid®; Etopophos®; VP-16; Etoposide phosphate
Drug: Cyclophosphamide, Thiotepa, Carboplatin (CTC) or STAMP V (CTC) — Cyclophosphamide will be given at a dose of 2000 mg/m2 in NS IV over one hour daily on days -4, -3, and -2 (total = 6000 mg/m2).
  Thiotepa will be given at a dose of 167 mg/m2 in NS IV over one hour daily on days -4, -3, -2 (total = 500 mg/m2) as the preparative regimen followed by PBSCT on day 0.
  Carboplatin will be given at a dose of 267 mg/m2 in D5W IV over one hour daily on days -4, -3, and -2.
  Mesna will be administered per BMT Standard of Care Guidelines at a dose of 25% of the total cyclophosphamide dose 30 minutes prior to and then 3, 6, and 9 hours after cyclophosphamide daily on days -4, -3, and -2 prior to PBSCT for a total of 2000mg/m2.
  Other Names: Cytoxan®; Neosar®; Paraplatin ®
Procedure: Leukapheresis — Peripheral blood mononuclear cells (PBMC) will be collected by leukapheresis (for generation of ATC) prior to or post G-CSF (16 ug/kg/day) priming for collecting stem cells.
Procedure: peripheral blood stem cell transplantation (PBSCT) — Will be collected either before or after peripheral blood stem cell collection for stem cell transplant.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation plus biological therapy may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: This phase II trial is studying how well chemotherapy followed by peripheral stem cell transplantation plus biological therapy works in treating women with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the use of autologous peripheral blood stem cell transplantation followed by immunotherapy with activated T cells in women with stage IV breast cancer improves progression-free survival (PFS) compared to a reported mean PFS in patients treated with second-line chemotherapy with matching inclusion criteria by published trials.
* Determine if this regimen improves clinical response and overall survival.
* Perform sequential immune monitoring studies, including phenotyping, cytotoxic assays, EliSpots for IFNγ, selected T-cell repertoire (Vβ analysis), HER2/new tetramer analysis, and serum tumor markers.
* Test correlations between immune function tests and clinical endpoints.

OUTLINE: Patients are stratified according to tumor classification (chemosensitive vs chemoresistant).

Patients receive filgrastim (G-CSF) subcutaneously (SC) daily for 4 days followed by peripheral blood mononuclear cell (PBMC) collection for PBSCT and generation of activated T cells (ATC). The PBMC are treated ex vivo with monoclonal antibody OKT3 to form ATC. The ATC are expanded for 12-14 days in interleukin-2 (IL-2).

Patients then receive high-dose chemotherapy. Patients with chemosensitive disease receive cyclophosphamide IV over 1 hour, thiotepa IV over 1 hour, and carboplatin IV over 1 hour on days -4, -3, and -2. Patients with chemoresistant disease receive ifosfamide IV over 1 hour, etoposide IV twice daily, and carboplatin IV over 1 hour on days -8 to -3. Patients undergo autologous PBSC transplantation on day 0 or on both day 0 and day 1.

Patients then receive ATC IV over 15-20 minutes three times per week starting approximately on day +1 for three weeks and then once weekly for at least 6 doses.

After completion of study therapy, patients are followed periodically for up to 2 years after PBSC.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Women with histologically documented metastatic carcinoma of the breast

  * Bilateral disease allowed
  * Concurrent intraductal or lobular carcinoma in situ allowed
* Measurable or evaluable recurrent metastatic disease (stage IV) documented by radiograph, CT scan, nuclear medicine scan, or physical exam

  * Biopsy of recurrent site(s) recommended but not required
  * Nonmeasurable disease allowed if tumor or metastatic disease has been previously removed or successfully treated
* 0 to 3+ HER2 amplification, as determined by FISH
* No clinical evidence of active brain metastases

  * Patients with treated brain metastases (i.e., those who have received definitive radiation, chemotherapy, and/or underwent surgery) and are stable are eligible
* Hormone receptor status:

  * Estrogen or progesterone receptor positive or negative

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Karnofsky performance status 70-100% OR ECOG performance status 0-2
* Life expectancy at least 3 months
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 50,000/mm^3
* Hemoglobin greater than 8 g/dL
* Bilirubin less than 1.5 times normal
* AST, ALT, and alkaline phosphatase < 5 times upper normal
* Creatinine less than 1.8 mg/dL
* Creatinine clearance at least 60 mL/min
* BUN less than 1.5 times normal
* No myocardial infarction (MI) within the past year
* No history of MI (> 1 year ago) with current coronary symptoms requiring medication
* No current history of angina/coronary symptoms requiring medication
* No clinical evidence of congestive heart failure requiring medical management
* No significant congestive heart failure
* No other uncontrolled or significant cardiovascular disease
* Ejection fraction at least 45% at rest by MUGA
* Systolic BP < 130 mm Hg and diastolic BP < 80 mm Hg

  * BP must be controlled to meet the standard by anti-hypertensive medications for at least 7 days prior to the first infusion
* PFT-FEV_1 at least 50% predicted
* DLCO2 at least 50% predicted
* FVC at least 50% predicted
* No other malignancy within the past 3 years
* No other serious medical or psychiatric illness that would preclude study participation
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior chemotherapy regimens allowed, including prior treatment on protocol WSU-2006-130
* Prior vaccine therapy on protocol WSU-2006-130 allowed
* More than 4 weeks to leukapheresis since prior hormonal therapy
* No radiation to the axial skeleton within 4 weeks of leukapheresis
* No concurrent hormonal therapy for breast cancer

  * Hormones administered for non-disease-related condition (e.g. insulin for diabetes) allowed
* Concurrent steroids for adrenal failure, septic shock, or pulmonary toxicity allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence G. Lum, MD, DSc, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Therapeutic Autologous Lymphocytes: therapeutic autologous lymphocytes: Immediately after pheresis.,The time for ATC infusions will vary from patient to patient, but the infusion rate will be approximately 10 × 109 ATC will be based on the rate calculated from the endotoxin level in the cell product. All patients will be observed for at least 1 hr after an infusion.
  Ifosfamide, carboplatin, and etoposide (ICE) regimen: Ifosfamide 2,500 mg/m2 given IV daily on day -8, -7, -6, -5, -4, and -3 prior to PBSCT. Ifosfamide 2,500 mg/m2 infused IV over 1 hour (hour 0-1) on days -8 to -3 for a total dose of 15,000 mg/m2.
  Mesna will be administered per BMT Standard of Care Guideline at a dose of 25% of the total Ifosfamide dose 30 minutes prior to and then 3, 6, and 9 hours after ifosfamide daily on days -8, -7, -6, -5, -4, and -3 prior to PBSCT for a total dose of 2500 m
Period: Overall Study
Arm/Group | Therapeutic Autologous Lymphocytes
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Therapeutic Autologous Lymphocytes: therapeutic autologous lymphocytes: Immediately after pheresis, the lymphocytes will be activated with soluble monoclonal anti-CD3 antibody (OKT3) which cross-links the CD3 receptors on T cells and activates T cells.
  The time for ATC infusions will vary from patient to patient, but the infusion rate will be approximately 10 × 109 ATC will be based on the rate calculated from the endotoxin level in the cell product. All patients will be observed for at least 1 hr after an infusion.
  Ifosfamide, carboplatin, and etoposide (ICE) regimen: Ifosfamide 2,500 mg/m2 given IV daily on day -8, -7, -6, -5, -4, and -3 prior to PBSCT. Ifosfamide 2,500 mg/m2 infused IV over 1 hour (hour 0-1) on days -8 to -3 for a total dose of 15,000 mg/m2.
  Mesna administered per BMT Standard of Care Guideline at a dose of 25% of the total Ifosfamide dose 30 mins. prior to and then 3, 6, and 9 hrs after ifosfamide daily on days -8, -7, -6, -5, -4, and -3 prior to PBSCT for a total dose of 2500 m
Arm/Group | Therapeutic Autologous Lymphocytes
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Time Frame: Length of time from day of transplant until recurrence or relapse.
Population: Trial converted to a proof-of-principle or concept trial; 7 eligible pts received their ATC infusions, 5 were evaluable. This small number of pts is not adequate for progression-free survival or overall survival analysis, collected and analyzed the data for cytotoxicity, IFN-g EliSpots and serum antibodies to monitor for immune responses.
Groups:
- Therapeutic Autologous Lymphocytes: therapeutic autologous lymphocytes: Immediately after pheresis.
  The time for ATC infusions will vary from patient to patient, but the infusion rate will be approximately 10 × 109 ATC will be based on the rate calculated from the endotoxin level in the cell product. All patients will be observed for at least 1 hr after an infusion.
  Ifosfamide, carboplatin, and etoposide (ICE) regimen: Ifosfamide 2,500 mg/m2 given IV daily on day -8, -7, -6, -5, -4, and -3 prior to PBSCT. Ifosfamide 2,500 mg/m2 infused IV over 1 hour (hour 0-1) on days -8 to -3 for a total dose of 15,000 mg/m2.
  Mesna will be administered per BMT Standard of Care Guideline at a dose of 25% of the total Ifosfamide dose 30 minutes prior to and then 3, 6, and 9 hours after ifosfamide daily on days -8, -7, -6, -5, -4, and -3 prior to PBSCT for a total dose of 2500 m
Arm/Group | Therapeutic Autologous Lymphocytes
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Time Frame: Length of time from day of transplant until death.
Population: as for outcome 1
Groups:
- Therapeutic Autologous Lymphocytes: therapeutic autologous lymphocytes: Immediately after pheresis, the lymphocytes will be activated with soluble monoclonal anti-CD3 antibody (OKT3) which cross-links the CD3 receptors on T cells and activates T cells.
  The time for ATC infusions will vary from patient to patient, but the infusion rate will be based on the rate calculated from the endotoxin level in the cell product. All patients will be observed for at least 1 hr after an infusion.
  Ifosfamide, carboplatin, and etoposide (ICE) regimen: Ifosfamide 2,500 mg/m2 given IV daily on day -8, -7, -6, -5, -4, and -3 prior to PBSCT. Ifosfamide 2,500 mg/m2 infused IV over 1 hour (hour 0-1) on days -8 to -3 for a total dose of 15,000 mg/m2.
  Mesna will be administered per BMT Standard of Care Guideline at a dose of 25% of the total Ifosfamide dose 30 minutes prior to and then 3, 6, and 9 hours after ifosfamide daily on days -8, -7, -6, -5, -4, and -3 prior to PBSCT for a total dose of 2500 mg/m2.
  Carboplatin at a dose of
Arm/Group | Therapeutic Autologous Lymphocytes
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Therapeutic Autologous Lymphocytes
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
Not enough funding to finish study, cost of immunotherapy infusions for the stem cell transplant portion & of infusions for targeted T cell therapy were limited due to lack of funding, trial was converted into a proof-of-principle or concept trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No